CLINICAL TRIAL: NCT03145987
Title: A Randomized, Double-blinded, Clinical Trial on Effects of a Food Supplement on Cognitive and Neuropsychological Functioning in Healthy Older Adults.
Brief Title: Effects of a Food Supplement on Cognitive and Neuropsychological Functioning in Older Adults.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Policlinico "G. Martino" (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PhCT-3
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Cognitive Decline; Neurophysiologic Abnormality
Keywords: Cognitive functioning; Neuropsychological status; Vitis vinifera
MeSH Terms: conditions — Cognitive Dysfunction | interventions — whole grape extract

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, placebo controlled study.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: subjects were randomly allocated to one of two groups treated as follows: Group 1, N = 57 to be treated with Cognigrape capsule (verum 250 mg/day); Group 2, N = 54 to be treated with placebo for 12 weeks. Neither subjects recruited for the study nor investigators knew the content of sachets or were able to differentiate the two different treatments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitis vinifera extract (Experimental): Vitis vinifera extract 250 mg/day orally administered for 12 weeks.
  Interventions: Dietary Supplement: Vitis vinifera extract
- Placebo (Placebo Comparator): Placebo orally administered once a day for 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitis vinifera extract
  Other Names: Cognigrape®
  Arms: Vitis vinifera extract
Other: Placebo
  Arms: Placebo

SUMMARY:
The increase in life expectancy is associated with a gradual aging of the population so creating new needs arising from this new situation. Memory ability declines with age and memory deficits are regarded as an initial symptom of dementia of Alzheimer's Disease (AD) type, one of the most prevalent cognitive disorders in older people. States and scientific community have been called to find preventive strategies acting against the consequent physiological cognitive decline with the aim to attenuate the increase of dementia. Numerous studies have shown that polyphenolic compounds derived from multiple dietary sources, and more specifically the polyphenolic compounds found in grapes (GP), are able to attenuate the cognitive impairment and in reducing neuropathological lesions in the brain in experimental animal models for the study of Alzheimer's Disease (AD) .

In recent years, several in vivo studies have shown that oral administration of polyphenols from grapes improves antioxidant status in the brain and prevents neuronal damage induced by free radicals. The intake of proanthocyanidins, especially in the monomeric form, showed to produce an improvement of cognitive function in an Alzheimer's disorder animal model.

A randomized, double-blind, placebo-controlled clinical trial was designed by the investigators with the aim to evaluate potential beneficial effects of a Vitis vinifera-based food supplement on cognitive functioning and neuropsychological status in healthy older adults aging 55-75 years.

For the enrollment, mental status was evaluated through the Mini-Mental State Exam, a test able to provide quickly a screen of orientation, providing a rapid screen of recall, language, orientation, registration, attention and calculation. 111 subjects were recruited and, after obtaining the informed consent, successively randomly divided in two groups: Group 1, N = 57 to be treated for 12 weeks with Vitis vinifera extract (verum 250 mg/day); Group 2, N = 54 to be treated for 12 weeks with placebo. Cognitive functioning and neuropsychological status were evaluated at the beginning (before treatment) and a the end of treatment by using Mini Mental State Examination (MMSE), Beck Depression Inventory (BDI), Hamilton Anxiety Rating Scale (HARS) and Repeatable Battery for the Assessment of Neuropsychological Status.

DETAILED DESCRIPTION:
Study design The study was a randomized into a two-group, parallel, placebo-controlled clinical trial to assess the efficacy of a food supplement containing vitis vinifera extract developed for cognitive and neuropsychological functioning in healthy older adults.

Screening Mental status was evaluated through the MMSE, a test able to provide quickly a screen of orientation, providing a rapid screen of recall, language, orientation, registration, attention and calculation. To study the effects on cognitive functioning and neuropsychological status participants were also subjected to the Beck Depression Inventory (BDI) and Hamilton Anxiety Rating Scale (HARS).

At screening (visit 1, day 0) after giving informed consent, subjects underwent medical history, physical examination, and vital signs. All subjects got oral and written information about the study and gave written informed consent to participate before inclusion in the trial. After screening and evaluation of baseline scores, included subjects were randomly allocated to one of two groups treated as follows: Group 1, N = 57 to be treated with Cognigrape capsule (verum 250 mg/day); Group 2, N = 54 to be treated with placebo . Randomisation by blocks of 3 (2 + 1) was double-blinded. Successive blocks were balanced by 2s. Neither subjects recruited for the study nor investigators were able to differentiate the two different treatments.

The Mini-Mental State Examination is composed of 12 items exploring through 22 trials verbal and performance, 7 cognitive functions: temporal and spatial orientation; immediate memory; attention and calculation; recall memory; language; praxia visuo-constructive. The administration requires a time ranging from 5 to 15 minutes. The score is corrected for age and education; the threshold for the purposes of enrollment in the study is set at a score ≥ 24. The MMSE score between 18 and 24 is an indication of a compromised moderate to mild, while a score of 25 is considered borderline, from 26 to 30 is indicative of normality cognitive. For this reason a score limit of 24 including masked potential light cognitive decline in healthy adults was chosen.

Beck Depression Inventory is a self-report instrument measuring the severity of depression. The Beck Depression Inventory (BDI) Short Form, a prominently and frequently cited, self-reported measure of depression was used. The 13-item questionnaire assesses 4 major components of depression: behavioral, affective, cognitive, and physiological. Numerical values assigned to each statement range from 0 to 3 indicating increasing severity. According to Beck's clinical criteria, a score between 8 and 15 indicates moderate depression and 16 severe depression.

Questionnaire is composed of in 21 questions with multiple choice response suitable to investigate the presence of depressive symptoms; aspects investigated by the test are: sadness, pessimism, sense of failure, dissatisfaction, guilty, free expectation, self-disappointment, self-accusation, suicidal ideas, crying, irritability, indecision, doubt, social withdrawal, devaluation of its image body, work efficiency decrease, sleep disturbance, fatigue, decreased appetite, weight loss, somatic concerns, loss of libido. The questionnaire has been administered immediately before the beginning (Day 0) and at the end of treatment (after 12 weeks).

Hamilton Anxiety Rating Scale is a scale evaluating anxiety through the investigation of 15 different areas (such as insomnia, mood, somatic symptoms). Each of the 15 areas is composed of a minimum of 3 to a maximum of 8 items to each of which is given a score from 0 to 6, depending on the severity of symptoms. Subsequently the total value is calculated for each area, using a score of 0 (absent), 1 (mild), 2 (moderate), 3 (severe), or 4 (very severe) points, based on the overall severity of symptoms investigating each specific area. The total score, which has been called "whole", is calculated by adding the points of each of the 15 areas surveyed. The rating of the scale may vary from 0 to 56. A total score around 18 is considered indicative of a pathological state.

Repeatable Battery for the Assessment of Neuropsychological Status is a quick and complete neuropsychological battery, consisting of two forms ( "A" and "B") associated with identical difficulty degrees, each divided into 12 subtests administered to evaluate 5 different cognitive domains: attention, language, visuospatial/constructional abilities immediate memory and delayed memory.

Cognitive-neuropsychological assessment was performed at baseline (o day) and after the 12 weeks of treatment period. Measures included MMSE, BDI, HARS, RBANS.

ELIGIBILITY:
Inclusion Criteria:

* age over 55 years; italian speaking and understanding; no using food supplements for cognitive functioning two weeks before enrolling and during the study period; score > or = 24 at Mini-Mental State Exam (MMSE).

Exclusion Criteria:

* age < 55 or > 75 years, or AD or other related disorders, psychiatric or neurological diseases (including aphasia, sensory, motor or visual disturbances which could affect the test results), cancer, coagulation disorders, cardiovascular, lung, kidney, thyroid, liver, gastrointestinal disease or insulin-dependent diabetes, excessive consumption of alcohol or substance abuse/dependence; more than 3 medical hospitalizations last year or subjects taking coumadin, tricyclic antidepressants, antipsychotics, and anticonvulsants or any medications for cognitive functioning.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Mini Mental State Examination | Up to 12 weeks
  Mini Mental state Examination is composed of 12 items exploring through 22 trials verbal and performance, 7 cognitive functions: temporal and spatial orientation; immediate memory; attention and calculation; recall memory; language; praxia visuo-constructive.
Beck Depression Inventory | Up to 12 weeks.
  It is a self-report instrument measuring the severity of depression. The Beck Depression Inventory (BDI) Short Form was used. BDI is a prominently and frequently cited, self-reported measure of depression. The 13-item questionnaire assesses 4 major components of depression: behavioral, affective, cognitive, and physiological. Numerical values assigned to each statement range from 0 to 3 indicating increasing severity. According to Beck's clinical criteria, a score between 8 and 15 indicates moderate depression and 16 severe depression.
Hamilton Anxiety Rating Scale | Up to 12 weeks.
  Hamilton Anxiety Rating Scale is a scale evaluating anxiety through the investigation of 15 different areas (such as insomnia, mood, somatic symptoms). Each of the 15 areas is composed of a minimum of 3 to a maximum of 8 items to each of which is given a score from 0 to 6, depending on the severity of symptoms. Subsequently the total value is calculated for each area, using a score of 0 (absent), 1 (mild), 2 (moderate), 3 (severe), or 4 (very severe) points, based on the overall severity of symptoms investigating each specific area. The total score, which has been called "whole", is calculated by adding the points of each of the 15 areas surveyed. The rating of the scale may vary from 0 to 56. A total score around 18 is considered indicative of a pathological state.
Repeatable Battery for the Assessment of Neuropsychological Status | Up to 12 weeks.
  Repeatable Battery for the Assessment of Neuropsychological Status is a quick and complete neuropsychological battery, consisting of two forms ( "A" and "B") associated with identical difficulty degrees, each divided into 12 subtests administered to evaluate 5 different cognitive domains: attention, language, visuospatial/constructional abilities immediate memory and delayed memory.

CONTACTS AND LOCATIONS:
Overall Officials: Umberto Alecci, MD, Principal Investigator — Azienda Ospedaliera Universitaria "G Martino", Messina, Italy.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andreescu C, Belnap BH, Rollman BL, Houck P, Ciliberti C, Mazumdar S, Shear MK, Lenze EJ. Generalized anxiety disorder severity scale validation in older adults. Am J Geriatr Psychiatry. 2008 Oct;16(10):813-8. doi: 10.1097/JGP.0b013e31817c6aab. PMID 18827227
- [Background] Asha Devi S, Sagar Chandrasekar BK, Manjula KR, Ishii N. Grape seed proanthocyanidin lowers brain oxidative stress in adult and middle-aged rats. Exp Gerontol. 2011 Nov;46(11):958-64. doi: 10.1016/j.exger.2011.08.006. Epub 2011 Aug 16. PMID 21871550
- [Background] Assuncao M, de Freitas V, Paula-Barbosa M. Grape seed flavanols, but not Port wine, prevent ethanol-induced neuronal lipofuscin formation. Brain Res. 2007 Jan 19;1129(1):72-80. doi: 10.1016/j.brainres.2006.10.044. Epub 2006 Dec 6. PMID 17156755
- [Background] Fremont L, Belguendouz L, Delpal S. Antioxidant activity of resveratrol and alcohol-free wine polyphenols related to LDL oxidation and polyunsaturated fatty acids. Life Sci. 1999;64(26):2511-21. doi: 10.1016/s0024-3205(99)00209-x. PMID 10403511
- [Background] He Q, Yang SY, Wang W, Wu ZJ, Ma HL, Lu Y. Proanthocyanidins affects the neurotoxicity of Abeta25-35 on C57/bl6 mice. Eur Rev Med Pharmacol Sci. 2016;20(4):679-84. PMID 26957270
- [Background] Oliboni LS, Dani C, Funchal C, Henriques JA, Salvador M. Hepatoprotective, cardioprotective, and renal-protective effects of organic and conventional grapevine leaf extracts on Wistar rat tissues. An Acad Bras Cienc. 2011 Dec;83(4):1403-11. doi: 10.1590/s0001-37652011000400027. PMID 22146965
- [Background] Shukitt-Hale B, Carey A, Simon L, Mark DA, Joseph JA. Effects of Concord grape juice on cognitive and motor deficits in aging. Nutrition. 2006 Mar;22(3):295-302. doi: 10.1016/j.nut.2005.07.016. Epub 2006 Jan 18. PMID 16412610
- [Background] Wang YJ, Thomas P, Zhong JH, Bi FF, Kosaraju S, Pollard A, Fenech M, Zhou XF. Consumption of grape seed extract prevents amyloid-beta deposition and attenuates inflammation in brain of an Alzheimer's disease mouse. Neurotox Res. 2009 Jan;15(1):3-14. doi: 10.1007/s12640-009-9000-x. Epub 2009 Feb 10. PMID 19384583
- [Background] Hartman RE, Shah A, Fagan AM, Schwetye KE, Parsadanian M, Schulman RN, Finn MB, Holtzman DM. Pomegranate juice decreases amyloid load and improves behavior in a mouse model of Alzheimer's disease. Neurobiol Dis. 2006 Dec;24(3):506-15. doi: 10.1016/j.nbd.2006.08.006. Epub 2006 Sep 28. PMID 17010630
- [Background] Hill NL, Mogle J, Wion R, Munoz E, DePasquale N, Yevchak AM, Parisi JM. Subjective Cognitive Impairment and Affective Symptoms: A Systematic Review. Gerontologist. 2016 Dec;56(6):e109-e127. doi: 10.1093/geront/gnw091. Epub 2016 Jun 23. PMID 27342440
- [Background] Novitski J, Steele S, Karantzoulis S, Randolph C. The Repeatable Battery for the Assessment of Neuropsychological Status effort scale. Arch Clin Neuropsychol. 2012 Mar;27(2):190-5. doi: 10.1093/arclin/acr119. Epub 2012 Jan 25. PMID 22277124
- [Background] Petersen RC, Doody R, Kurz A, Mohs RC, Morris JC, Rabins PV, Ritchie K, Rossor M, Thal L, Winblad B. Current concepts in mild cognitive impairment. Arch Neurol. 2001 Dec;58(12):1985-92. doi: 10.1001/archneur.58.12.1985. PMID 11735772
- [Background] Randolph C, Tierney MC, Mohr E, Chase TN. The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS): preliminary clinical validity. J Clin Exp Neuropsychol. 1998 Jun;20(3):310-9. doi: 10.1076/jcen.20.3.310.823. PMID 9845158
- [Background] Rezai-Zadeh K, Shytle D, Sun N, Mori T, Hou H, Jeanniton D, Ehrhart J, Townsend K, Zeng J, Morgan D, Hardy J, Town T, Tan J. Green tea epigallocatechin-3-gallate (EGCG) modulates amyloid precursor protein cleavage and reduces cerebral amyloidosis in Alzheimer transgenic mice. J Neurosci. 2005 Sep 21;25(38):8807-14. doi: 10.1523/JNEUROSCI.1521-05.2005. PMID 16177050
- [Background] Scola G, Conte D, Spada PW, Dani C, Vanderlinde R, Funchal C, Salvador M. Flavan-3-ol compounds from wine wastes with in vitro and in vivo antioxidant activity. Nutrients. 2010 Oct;2(10):1048-59. doi: 10.3390/nu2101048. Epub 2010 Oct 11. PMID 22253995
- [Background] Seidel S, Dal-Bianco P, Pablik E, Muller N, Schadenhofer C, Lamm C, Klosch G, Moser D, Klug S, Pusswald G, Auff E, Lehrner J. Depressive Symptoms are the Main Predictor for Subjective Sleep Quality in Patients with Mild Cognitive Impairment--A Controlled Study. PLoS One. 2015 Jun 19;10(6):e0128139. doi: 10.1371/journal.pone.0128139. eCollection 2015. PMID 26090659
- [Background] Wang J, Ferruzzi MG, Ho L, Blount J, Janle EM, Gong B, Pan Y, Gowda GA, Raftery D, Arrieta-Cruz I, Sharma V, Cooper B, Lobo J, Simon JE, Zhang C, Cheng A, Qian X, Ono K, Teplow DB, Pavlides C, Dixon RA, Pasinetti GM. Brain-targeted proanthocyanidin metabolites for Alzheimer's disease treatment. J Neurosci. 2012 Apr 11;32(15):5144-50. doi: 10.1523/JNEUROSCI.6437-11.2012. PMID 22496560
- [Background] Wang J, Ho L, Zhao W, Ono K, Rosensweig C, Chen L, Humala N, Teplow DB, Pasinetti GM. Grape-derived polyphenolics prevent Abeta oligomerization and attenuate cognitive deterioration in a mouse model of Alzheimer's disease. J Neurosci. 2008 Jun 18;28(25):6388-92. doi: 10.1523/JNEUROSCI.0364-08.2008. PMID 18562609
- [Background] Vecchio F, Miraglia F, Quaranta D, Granata G, Romanello R, Marra C, Bramanti P, Rossini PM. Cortical connectivity and memory performance in cognitive decline: A study via graph theory from EEG data. Neuroscience. 2016 Mar 1;316:143-50. doi: 10.1016/j.neuroscience.2015.12.036. Epub 2015 Dec 24. PMID 26724581
- [Background] Studer J, Donati A, Popp J, von Gunten A. Subjective cognitive decline in patients with mild cognitive impairment and healthy older adults: association with personality traits. Geriatr Gerontol Int. 2014 Jul;14(3):589-95. doi: 10.1111/ggi.12139. Epub 2013 Aug 29. PMID 23992484
- [Background] Small GW, Chen ST, Komo S, Ercoli L, Miller K, Siddarth P, Kaplan A, Dorsey D, Lavretsky H, Saxena S, Bookheimer SY. Memory self-appraisal and depressive symptoms in people at genetic risk for Alzheimer's disease. Int J Geriatr Psychiatry. 2001 Nov;16(11):1071-7. doi: 10.1002/gps.481. PMID 11746653